CLINICAL TRIAL: NCT03360539
Title: Nurse-Family Partnership Impact Evaluation in South Carolina
Acronym: NFP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Abdul Latif Jameel Poverty Action Lab (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, Margaret McConnell, Associate Professor of Global Health Economics, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB15-2939
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Preterm Birth; Injuries; Maternal Behavior
MeSH Terms: conditions — Premature Birth; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The Nurse-Family Partnership (NFP) was launched by pediatrician David Olds in the early 1970s in response to the observation that low-income mothers are less likely to engage in positive health and parenting behaviors that are associated with better child development outcomes (Olds et al. 1986). NFP is a prenatal and infancy home visiting program for low-income, first-time mothers and their families. Registered nurses begin visiting their clients as early in the pregnancy as possible, helping the mother-to-be make informed choices. The nurses continue visiting regularly until the child is two years old.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment-NFP (Experimental): NFP is a prenatal and infancy home visiting program for low-income, first-time mothers and their families. Registered nurses begin visiting their clients as early in the pregnancy as possible, helping the mother-to-be make informed choices. The nurses continue visiting regularly until the child is two years old.
  Interventions: Behavioral: Nurse-Family Partnership
- Control (No Intervention): Control group members have access to the standard of care and whatever other programs and services are available in the community.

INTERVENTIONS:
Behavioral: Nurse-Family Partnership
  Arms: Treatment-NFP

SUMMARY:
This study evaluates the effects of the Nurse Family Partnership (NFP), an established home-visiting program, using a scientifically rigorous individual-level randomized controlled trial. The study will be based in South Carolina, where a Medicaid waiver in combination with a pay-for-success contract will allow expansion of the program to women on Medicaid. The study plans to enroll 4000 low-income, first time mothers and their children into the intervention group, and another 2000 into the control group. The study will evaluate the program's impacts on outcomes using administrative records. This study aims to yield new evidence on the effect of NFP in a modern context, applied to a new population, across a broad range of outcomes, and financed by a novel public-private partnership based on accountability for outcomes.

DETAILED DESCRIPTION:
This study is an individual-level randomized controlled trial, with randomization post-consent. The study will enroll pregnant women who are income-eligible for Medicaid, less than 28 weeks pregnant, and have not had a previous live birth. All eligible applicants who provide written consent will be randomly assigned either to a treatment group that is offered access to NFP or to a control group that is not. Two-thirds of those recruited will be randomized to the treatment group and one-third to the control group. Control group members will have access to the standard of care and whatever other programs and services are available in the community.

The investigators will assess the effect of NFP on a range of short- and long-run maternal and child outcomes using administrative data that will be available for all members of both treatment and control groups. Several of the outcomes the investigators will evaluate are required as part of the Medicaid waiver and pay-for-success financing model.

ELIGIBILITY:
Inclusion Criteria:

* Female
* No previous live births
* Currently pregnant
* Gestation period less than 28 weeks (i.e. less than or equal to 27 weeks, 6 days) at time of recruitment
* Ages 15-55
* Income level meets Medicaid eligibility criteria
* Live within an area serviced by a NFP Implementing Agency
* Not currently enrolled in the study
* Not incarcerated or living in lock down facilities

Exclusion Criteria:

* Men
* Women who have had a previous live birth
* Women who are not currently pregnant
* Women who are past their 28th week of gestation (i.e. greater than or equal to 28 weeks, 0 days) at time of recruitment
* Women who are younger than 15 or older than 55 years of age
* Women whose income level does not meet Medicaid eligibility criteria
* Women who live outside of an area serviced by a NFP Implementing Agency
* Women who are currently enrolled in the study
* Women who are currently incarcerated or living in a lock down facility

Ages: 15 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5670 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2046-04-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret McConnell, PhD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (9):
- United States (9):
  - Nurse-Family Partnership of Anderson County, Anderson, South Carolina
  - NFP of Berkeley/Charleston/Dorchester Counties, Charleston, South Carolina
  - Nurse-Family Partnership of Lexington-Richland Co., Columbia, South Carolina
  - Nurse-Family Partnership of Horry County, Conway, South Carolina
  - McLeod Health NFP, Florence, South Carolina
  - Nurse-Family Partnership of Greenville County, Greenville, South Carolina
  - Carolina Health Centers NFP, Greenwood, South Carolina
  - Family Solutions of the Lowcountry NFP, Orangeburg, South Carolina
  - Spartanburg Regional Hospital NFP, Spartanburg, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swanson K, Ayers S, Oviedo D, Zhou RA, Bates MA, Baicker K, Chien AT, McConnell M. Intensive Nurse Home Visiting and Early Childhood Outcomes: A Randomized Clinical Trial. JAMA Pediatr. 2025 Aug 1;179(8):857-866. doi: 10.1001/jamapediatrics.2025.1600. PMID 40522648
- [Derived] Rokicki S, Oviedo D, Perreault N, Bates MA, Zhou RA, Baicker K, McConnell MA. Impact of nurse home visiting on take-up of social safety net programs in a Medicaid population. Health Aff Sch. 2025 Apr 2;3(4):qxaf038. doi: 10.1093/haschl/qxaf038. eCollection 2025 Apr. PMID 40177469
- [Derived] Rokicki S, Oviedo D, Perreault N, Zera C, McGregor AJ, Bates MA, Zhou RA, Baicker K, McConnell MA. Home Visits and the Use of Routine and Emergency Postpartum Care Among Low-Income People: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Dec 2;7(12):e2451605. doi: 10.1001/jamanetworkopen.2024.51605. PMID 39714843
- [Derived] Steenland MW, Oviedo D, Bates MA, Zhou A, Zera C, Baicker K, McConnell MA. Effect of an Intensive Nurse Home Visiting Program on Postpartum Contraceptive Use and Birth Spacing: A Randomized Controlled Trial. Obstet Gynecol. 2025 Jan 1;145(1):3-12. doi: 10.1097/AOG.0000000000005786. Epub 2024 Nov 14. PMID 39671266
- [Derived] McConnell MA, Rokicki S, Ayers S, Allouch F, Perreault N, Gourevitch RA, Martin MW, Zhou RA, Zera C, Hacker MR, Chien A, Bates MA, Baicker K. Effect of an Intensive Nurse Home Visiting Program on Adverse Birth Outcomes in a Medicaid-Eligible Population: A Randomized Clinical Trial. JAMA. 2022 Jul 5;328(1):27-37. doi: 10.1001/jama.2022.9703. PMID 35788794
- [Derived] McConnell MA, Zhou RA, Martin MW, Gourevitch RA, Steenland M, Bates MA, Zera C, Hacker M, Chien A, Baicker K. Protocol for a randomized controlled trial evaluating the impact of the Nurse-Family Partnership's home visiting program in South Carolina on maternal and child health outcomes. Trials. 2020 Dec 4;21(1):997. doi: 10.1186/s13063-020-04916-9. PMID 33276816

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment - Participation in Nurse Family Partnership: NFP is a prenatal and infancy home visiting program for low-income, first-time mothers and their families. Registered nurses begin visiting their clients as early in the pregnancy as possible, helping the mother-to-be make informed choices. The nurses continue visiting regularly until the child is two years old.
Period: Overall Study
Arm/Group | Treatment - Participation in Nurse Family Partnership | Control
Started | 3806 | 1864
Participants matched to index birth or index fetal death (Participants who experienced an index fetal death are excluded from most outcome analyses except where otherwise noted.) | 3319 | 1647
Completed | 3295 | 1637
Not Completed | 511 | 227

BASELINE CHARACTERISTICS:
Population: The total number of participants in the baseline analysis includes randomized participants who were successfully matched to an index birth or fetal death and excludes those who were not. This sample also excludes participants who withdrew from the study, experienced a pregnancy loss/miscarriage, or who did not receive the treatment as assigned.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment - Participation in Nurse Family Partnership | Control | Total
Number analyzed (Participants) | 3319 | 1647 | 4966
Age, Customized [Count of Participants; unit: Participants]
  Age in years: 15-18 years | 605 | 290 | 895
  Age in years: 19-24 | 1814 | 905 | 2719
  Age in years: 25-34 | 806 | 418 | 1224
  Age in years: 35+ | 94 | 34 | 128
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3319 | 1647 | 4966
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Row population differs due to missing/non-reported values.
  Participants
    Race and Ethnicity: number analyzed (Participants) | 3118 | 1530 | 4648
    Race and Ethnicity: Asian, Indigenous, Native Hawaiian and Pacific Islander, non-Hispanic | 44 | 12 | 56
    Race and Ethnicity: Hispanic | 173 | 95 | 268
    Race and Ethnicity: More than once race reported, non-Hispanic | 97 | 45 | 142
    Race and Ethnicity: Non-Hispanic Black | 1713 | 852 | 2565
    Race and Ethnicity: Non-Hispanic White | 1091 | 526 | 1617
Region of Enrollment [Number; unit: participants]
  United States | 3319 | 1647 | 4966
Highest education level [Count of Participants; unit: Participants] — Population: Row population differs due to missing/non-reported values.
  Participants
    number analyzed (Participants) | 3305 | 1641 | 4946
    Less than high school diploma | 750 | 358 | 1108
    High school diploma or equivalent | 1187 | 561 | 1748
    Some college, less than bachelor's degree | 1121 | 592 | 1713
    Bachelor's degree or higher | 247 | 130 | 377
Economic conditions at time of enrollment [Count of Participants; unit: Participants] — Population: Row population differs due to missing/non-reported values.
  Participants
    Received at least one social service program: number analyzed (Participants) | 3255 | 1610 | 4865
    Received at least one social service program | 2133 | 1076 | 3209
    Worked for pay: number analyzed (Participants) | 3318 | 1646 | 4964
    Worked for pay | 1753 | 867 | 2620
    Lived with parents: number analyzed (Participants) | 3317 | 1645 | 4962
    Lived with parents | 1439 | 729 | 2168
    Experienced housing insecurity: number analyzed (Participants) | 3314 | 1643 | 4957
    Experienced housing insecurity | 549 | 287 | 836
Received mental health treatment in last year [Count of Participants; unit: Participants] — Population: Row population differs due to missing/non-reported values.
  Participants
    number analyzed (Participants) | 3316 | 221 | 3537
    (all) | 458 | 221 | 679
High stress [Count of Participants; unit: Participants] — Defined as a Perceived Stress Scale 4 (PSS-4) score ≥ 4. Based on the total score, which ranges from 0-16, with higher values indicating more severe stress. Population: Row population differs due to missing/non-reported values.
  Participants
    number analyzed (Participants) | 3274 | 1625 | 4899
    (all) | 2161 | 1073 | 3234
Depressive symptoms [Count of Participants; unit: Participants] — Defined as a Patient Health Questionnaire-2 score ≥ 3. Based on the total score, which ranges from 0-6, with higher values indicating more severe symptoms of depression. Population: Row population differs due to missing/non-reported values.
  Participants
    number analyzed (Participants) | 3294 | 1641 | 4935
    (all) | 635 | 305 | 940

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Composite Birth Outcome
Description: Composite of at least one of: small for gestational (SGA), or low birth weight (LBW) less than 2500 grams, preterm birth (PTB) less than 37 weeks' gestation (obstetric estimate), or perinatal mortality (fetal death at or after 20 weeks of gestation or mortality in the first 7 days of life).
Time Frame: 0-7 days after index birth; vital records, mortality records, and fetal death records
Population: Differs from randomized sample as it excludes participants who withdrew, who experienced a pregnancy loss, and who could not be matched to an index pregnancy.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership: NFP is a prenatal and infancy home visiting program for low-income, first-time mothers and their families. Registered nurses begin visiting their clients as early in the pregnancy as possible, helping the mother-to-be make informed choices. The nurses continue visiting regularly until the child is two years old.
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3319 | 1647
Participants | 892 | 430
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.5, 95% CI 2-sided [-2.1 to 3.1] — Adjusted between-group difference in the percentage of participants

2. Primary Outcome: Number of Participants Whose Child Experienced a Major Injury or Concern for Abuse or Neglect
Description: Composite of at least one health care encounter or mortality associated with International Classification of Diseases (ICD) codes indicating either major injury, or, concern for abuse or neglect for the participant's index child(ren).
Time Frame: within 24 months after index birth; Medicaid claims or hospital discharge data
Population: Differs from randomized sample as it excludes participants with an index fetal death, who withdrew, who experienced a pregnancy loss, and who could not be matched to an index pregnancy.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 901 | 438
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.4, 95% CI 2-sided [-2.3 to 3.0] — Adjusted between-group difference in the percentage of participants

3. Primary Outcome: Number of Participants With an Inter-birth Interval of < 21 Months
Description: Having a subsequent birth within the first 21 months of the index birth
Time Frame: within 21 months after index birth; vital records
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 363 | 199
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -1.1, 95% CI 2-sided [-2.9 to 0.8] — Adjusted between-group difference in the percentage of participants

4. Secondary Outcome: Number of Participants With an Infant Born Small for Gestational Age (SGA)
Description: Infant birth weight below the 10th percentile for infants of the same gestational age
Time Frame: At index birth; vital records
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 553 | 265
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.7, 95% CI 2-sided [-1.5 to 2.9] — Adjusted between-group difference in the percentage of participants

5. Secondary Outcome: Number of Participants With an Infant Born Large for Gestational Age (LGA)
Description: Infant birth weight above the 90th percentile for infants of the same gestational age
Time Frame: At index birth birth; vital records
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 166 | 95
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -0.9, 95% CI 2-sided [-2.3 to 0.4] — Adjusted between-group difference in the percentage of participants

6. Secondary Outcome: Number of Participants With an Infant Born With Low Birth Weight (LBW)
Description: Number of participants with an infant born with a birth weight of less than 2500 grams.
Time Frame: At index birth; vital records
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 436 | 219
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -0.4, 95% CI 2-sided [-2.4 to 1.6] — Adjusted between-group difference in the percentage of participants

7. Secondary Outcome: Number of Participants With an Infant With Very Low Birth Weight
Description: Number of participants with an infant born with a birth weight of less than 1500 grams.
Time Frame: At index birth; vital records
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 78 | 48
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -0.7, 95% CI 2-sided [-1.6 to 0.3] — Adjusted between-group difference in the percentage of participants

8. Secondary Outcome: Birth Weight (Continuous)
Description: A continuous measure of infant birth weight (grams)
Time Frame: At index birth; vital records
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
grams | 3085.2 (609.6) | 3095.7 (38.1)
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -7.8, 95% CI 2-sided [-43.7 to 28.0] — Adjusted between-group difference, in grams

9. Secondary Outcome: Number of Participants With a Preterm Birth
Description: Infant born before 37 weeks' gestation (obstetric estimate)
Time Frame: At index birth; vital records
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 379 | 190
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -0.5, 95% CI 2-sided [-2.4 to 1.3] — Adjusted between-group difference in the percentage of participants

10. Secondary Outcome: Number of Participants With an Extremely Preterm Birth
Description: Number of participants with an infant born before 28 weeks' gestation.
Time Frame: At index birth; vital records
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 32 | 16
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.0, 95% CI 2-sided [-0.6 to 0.5] — Adjusted between-group difference in the percentage of participants

11. Secondary Outcome: Gestational Age at Birth
Description: Gestational age at birth in weeks (continuous)
Time Frame: At index birth; vital records
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
weeks | 38.2 (2.3) | 38.1 (2.3)
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.1, 95% CI 2-sided [0.0 to 0.2] — Adjusted between-group difference, in weeks

12. Secondary Outcome: Number of Participants Experiencing Perinatal Mortality
Description: Fetal death at or after 20 weeks of gestation or mortality in the first 7 days of life
Time Frame: Within 1 week after index birth; mortality records and fetal death records
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3319 | 1647
Participants | 27 | 10
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.3, 95% CI 2-sided [-0.3 to 0.8] — Adjusted between-group difference in the percentage of participants

13. Secondary Outcome: Number of Participants With a NICU Admission of at Least Overnight
Description: Infant admitted to the neonatal intensive care unit (NICU) for at least one night
Time Frame: At index birth; hospital discharge
Population: Differs from randomized sample as it excludes participants with missing outcome data, those who experienced an index fetal death, who withdrew, who experienced a pregnancy loss, and who could not be matched to an index pregnancy.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3046 | 1497
Participants | 241 | 128
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -0.8, 95% CI 2-sided [-2.5 to 0.9] — Adjusted between-group difference in the percentage of participants

14. Secondary Outcome: Number of Participants Experiencing Neonatal Morbidity
Description: Assisted ventilation immediately after delivery, assisted ventilation for more than six hours, seizure, receipt of surfactant replacement therapy, and receipt of antibiotics for suspected sepsis.
Time Frame: At index birth; hospital discharge
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1647
Participants | 328 | 144
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.7, 95% CI 2-sided [-1.1 to 2.4] — Adjusted between-group difference in the percentage of participants

15. Secondary Outcome: Number of Participants Experiencing Cesarean Delivery
Description: Number of participants experiencing a cesarean delivery for their index birth.
Time Frame: At index birth; vital records
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 1015 | 530
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -2.0, 95% CI 2-sided [-4.7 to 0.7] — Adjusted between-group difference in the percentage of participants

16. Secondary Outcome: Number of Participants Experiencing Severe Acute Maternal Morbidity
Description: Severe acute maternal morbidity as defined by the Centers for Disease Control and Prevention (CDC).
Time Frame: At index birth; hospital discharge
Population: The analysis population for this outcome includes participants who matched to an index birth in claims data.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3464 | 1694
Participants | 56 | 23
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.2, 95% CI 2-sided [-0.5 to 0.9] — Adjusted between-group difference in the percentage of participants

17. Secondary Outcome: Number of Participants Experiencing Maternal Mortality
Description: Number of participants experiencing all-cause mortality within one year postpartum.
Time Frame: Within one year after index birth; mortality records
Population: Differs from randomized sample as it excludes participants with missing outcome data, an index fetal death, who withdrew, who experienced a pregnancy loss, and who could not be matched to an index pregnancy.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 5 | 1

18. Secondary Outcome: Number of Participants Experiencing Neonatal Abstinence Disorder (NAS) or Maternal Drug/Substance Abuse
Description: Number of participants experiencing neonatal abstinence disorder (NAS) or maternal drug/substance abuse in the first two years postpartum.
Time Frame: Within two years after index birth; Medicaid claims, hospital discharge
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 708 | 367

19. Secondary Outcome: Number of Participants Experiencing Violence or Homicide
Description: Includes any ICD code for healthcare encounter associated with experiencing violence or mortality associated with homicide based on ICD code
Time Frame: Within 2 years after index birth; Medicaid claims, mortality records
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 55 | 27

20. Secondary Outcome: Number of Participants With a Postpartum Visit
Description: Number of participants with a postpartum visit in first 12 weeks after an index birth.
Time Frame: Within 12 weeks after index birth; Medicaid claims
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3261 | 1616
Participants | 2079 | 1038
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -0.3, 95% CI 2-sided [-3.2 to 2.5] — Adjusted between-group difference in the percentage of participants

21. Secondary Outcome: Number of Participants Who Received Adequate Prenatal Care
Description: With adequacy defined using the Adequacy of Prenatal Care Utilization Index (APNCU), where prenatal care began by the 4th month and at least 80% of recommended visits were attended
Time Frame: At index birth; vital records
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership | Control
Number analyzed (Participants) | 3065 | 1522
Participants | 2572 | 1283
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -0.66, 95% CI 2-sided [-3.0 to 1.7] — Adjusted between-group difference in the percentage of participants

22. Secondary Outcome: Number of Emergency Department Visits During Pregnancy
Description: Number of emergency department visits during pregnancy.
Time Frame: At index birth; hospital discharge
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Treatment - Participation in Nurse Family Partnership | Control
Number analyzed (Participants) | 3065 | 1522
number of visits | 2.1 (2.5) | 2.0 (2.5)
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 1.01, 95% CI 2-sided [0.95 to 1.08] — Adjusted between-group difference, in number of visits

23. Secondary Outcome: Number of Participants With a Dental Visit During Pregnancy
Description: Number of participants with a dental visit during pregnancy (preventive or treatment).
Time Frame: At index birth; Medicaid claims and dental records
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership | Control
Number analyzed (Participants) | 3065 | 1522
Participants | 625 | 275
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 2.47, 95% CI 2-sided [0.1 to 4.9] — Adjusted between-group difference in the percentage of participants

24. Secondary Outcome: Number of Participants With an Ultrasound at 18-22 Weeks
Description: Number of participants with an ultrasound (anatomy scan) at 18-22 weeks.
Time Frame: 18-22 weeks gestation during index pregnancy. Assessed at index birth using Medicaid claims.
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership | Control
Number analyzed (Participants) | 3065 | 1522
Participants | 2293 | 1134
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.44, 95% CI 2-sided [-2.1 to 3.0] — Adjusted between-group difference in the percentage of participants

25. Secondary Outcome: Number of Participants Who Received Prenatal Screens
Description: Our original prenatal screening outcome variable included the obstetric panel: Rhesus-D (DRh), red blood cell (RBC) antibody screen, complete blood count (CBC), urine culture, urinalysis; sexually transmitted infection (STI) screenings (HIV, syphilis, hepatitis B, chlamydia if <25, gonorrhea if <25); Group B strep screening, and glucose screening. However, since most participants had already completed their first prenatal visit prior to enrolling in the trial (when many of these tests are performed), it was not appropriate to include first-visit tests as outcomes. We therefore modified the outcome to instead use three clinically relevant measures that could occur after enrollment: glucose screening, Group B strep screening, and Tdap vaccination. These outcomes are reported as they appear in the published papers.
Time Frame: At index birth; Medicaid claims
Reporting Status: Not Posted

26. Secondary Outcome: Number of Participants Who Received a Gestational Diabetes Test (24-28 Weeks)
Description: Received a glucose screen at 24-28 weeks' gestation.
  Note: Our original prenatal screening outcome variable included the obstetric panel (D [Rh], RBC antibody screen, CBC, urine culture, urinalysis), STI screenings (HIV, syphilis, hepatitis B, chlamydia if <25, gonorrhea if <25), Group B strep screening, and glucose screening. However, since most participants had already completed their first prenatal visit prior to enrolling in the trial (when many of these tests are performed), it was not appropriate to include first-visit tests as outcomes. We therefore modified the outcome to instead use three clinically relevant measures that could occur after enrollment: glucose screening, Group B strep screening, and Tdap vaccination. These outcomes are reported as they appear in the published papers.
Time Frame: At 24-28 weeks' gestation of index pregnancy; Medicaid claims
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership | Control
Number analyzed (Participants) | 3028 | 1502
Participants | 1747 | 869
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -0.12, 95% CI 2-sided [-3.1 to 2.9] — Adjusted between-group difference in the percentage of participants

27. Secondary Outcome: Number of Participants With a Tdap Vaccination (27-36 Weeks)
Description: Received Tdap vaccination at 27-36 weeks' gestation.
  Our original prenatal screening outcome variable included the obstetric panel (D [Rh], RBC antibody screen, CBC, urine culture, urinalysis), STI screenings (HIV, syphilis, hepatitis B, chlamydia if <25, gonorrhea if <25), Group B strep screening, and glucose screening. However, since most participants had already completed their first prenatal visit prior to enrolling in the trial (when many of these tests are performed), it was not appropriate to include first-visit tests as outcomes. We therefore modified the outcome to instead use three clinically relevant measures that could occur after enrollment: glucose screening, Group B strep screening, and Tdap vaccination. These outcomes are reported as they appear in the published papers.
Time Frame: At 27-36 weeks' gestation of index pregnancy; Medicaid claims
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership | Control
Number analyzed (Participants) | 2723 | 1347
Participants | 914 | 446
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.65, 95% CI 2-sided [-2.4 to 3.7] — Adjusted between-group difference in the percentage of participants

28. Secondary Outcome: Number of Participants With a Group B Streptococcus Test (35-37 Weeks)
Description: Received Group B streptococcus test at 35-37 weeks' gestation.
  Note: Our original prenatal screening outcome variable included the obstetric panel (D [Rh], RBC antibody screen, CBC, urine culture, urinalysis), STI screenings (HIV, syphilis, hepatitis B, chlamydia if <25, gonorrhea if <25), Group B strep screening, and glucose screening. However, since most participants had already completed their first prenatal visit prior to enrolling in the trial (when many of these tests are performed), it was not appropriate to include first-visit tests as outcomes. We therefore modified the outcome to instead use three clinically relevant measures that could occur after enrollment: glucose screening, Group B strep screening, and Tdap vaccination. These outcomes are reported as they appear in the published papers.
Time Frame: At 35-37 weeks' gestation of index pregnancy; Medicaid claims
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership | Control
Number analyzed (Participants) | 1807 | 885
Participants | 1150 | 602
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -4.18, 95% CI 2-sided [-8.0 to -0.4] — Adjusted between-group difference in the percentage of participants

29. Secondary Outcome: Number of Participants With a Mental Health Diagnosis or Outpatient Treatment
Description: Diagnosis for depression/anxiety/stress reaction or antidepressant prescription or outpatient mental health visit
Time Frame: During index pregnancy or 60 days postpartum; Medicaid claims
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 1048 | 543

30. Secondary Outcome: Number of Participants With a Diagnosis of Depression/Anxiety/Stress Reaction
Description: Number of participants with a diagnosis of depression/anxiety/stress reaction.
Time Frame: During index pregnancy or 60 days postpartum; Medicaid claims
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 937 | 491

31. Secondary Outcome: Number of Participants With an Antidepressant Prescription
Description: Number of participants with an antidepressant prescription.
Time Frame: During index pregnancy or 60 days postpartum; Medicaid claims
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 435 | 216

32. Secondary Outcome: Number of Participants With an Outpatient Mental Health Visit
Description: Number of participants with at least one outpatient mental health visit.
Time Frame: During index pregnancy or 60 days postpartum; Medicaid claims
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 165 | 76

33. Secondary Outcome: Number of Participants With a Mental Health Treatment Follow up
Description: Second antidepressant prescription or outpatient mental health visit within 120 days of treatment initiation ("acute phase")
Time Frame: Within 120 days of treatment initiation; Medicaid claims
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 292 | 142

34. Secondary Outcome: Number of Participants With a Mental Health Related Emergency/Inpatient Visit
Description: Based on all-listed diagnoses (i.e. primary or secondary) for depression/anxiety/stress reaction
Time Frame: During index pregnancy or 12 months postpartum; Hospital discharge
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 459 | 202

35. Secondary Outcome: Number of Mental Health Related Emergency/Inpatient Visits
Description: Based on all-listed diagnoses (i.e. primary or secondary) for depression/anxiety/stress reaction
Time Frame: During index pregnancy or 12 months postpartum; Hospital discharge
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
number of visits | .24 (0.89) | .21 (0.83)

36. Secondary Outcome: Number of Participants Whose Child Experienced a Major Injury
Description: Health care encounter or mortality associated with ICD codes indicating major injury
Time Frame: Within 24 months after index birth; Medicaid claims, hospital discharge, mortality records
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 878 | 430
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.2, 95% CI 2-sided [-2.4 to 2.8] — Adjusted between-group difference in the percentage of participants

37. Secondary Outcome: Number of Participants Whose Child Experienced Concern for Abuse or Neglect
Description: Health care encounter or mortality associated with ICD codes indicating concern for abuse or neglect
Time Frame: Within 24 months after index birth; Medicaid claims, hospital discharge, mortality records
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 137 | 66
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.1, 95% CI 2-sided [-1.1 to 1.3] — Adjusted between-group difference in the percentage of participants

38. Secondary Outcome: Number of Injuries
Description: Number of injuries for child
Time Frame: Within 24 months after index birth; hospital discharge
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of injuries
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
number of injuries | 0.2 (0.6) | 0.3 (0.6)
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.0, 95% CI 2-sided [-0.1 to 0.1] — Adjusted between-group difference, in number of injuries

39. Secondary Outcome: Number of Participants Whose Child Had an Emergency Department Visit
Description: Number of participants whose child had at least one visit to the emergency department.
Time Frame: Within 24 months after index birth; hospital discharge
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 2306 | 1192
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -2.7, 95% CI 2-sided [-5.3 to -0.1] — Adjusted between-group difference in the percentage of participants

40. Secondary Outcome: Number of Child Emergency Department Visits
Description: Total number of child visits to the emergency department (without admission)
Time Frame: Within 24 months after index birth; hospital discharge
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
number of visits | 2.3 (2.8) | 2.4 (2.8)
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -0.3, 95% CI 2-sided [-0.7 to 0.1] — Adjusted between-group difference, in number of visits

41. Secondary Outcome: Number of Participants Experiencing Child Mortality
Description: All-cause child mortality in first 24 months of life
Time Frame: Within 24 months after index birth; Mortality records
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3319 | 1647
Participants | 49 | 21
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.3, 95% CI 2-sided [-0.4 to 1.0] — Adjusted between-group difference in the percentage of participants

42. Secondary Outcome: Number of Participants With Recommended Number of Well-child Visits
Description: Number of participants that received the recommended number of well-child visits.
Time Frame: At 15 months after index birth; Medicaid claims
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 1150 | 537
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 2.3, 95% CI 2-sided [-0.4 to 5.0] — Adjusted between-group difference in the percentage of participants

43. Secondary Outcome: Number of Participants With Lead Screening
Description: Number of participants whose child received at least one lead screening.
Time Frame: At 15 months after index birth; Medicaid claims
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 2093 | 1030
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.5, 95% CI 2-sided [-2.3 to 3.2] — Adjusted between-group difference in the percentage of participants

44. Secondary Outcome: Number of Participants With Developmental Screening
Description: Number of participants whose child received at least one developmental screening.
Time Frame: At 12 months after index birth; Medicaid claims
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 1070 | 540
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -0.7, 95% CI 2-sided [-3.4 to 2.0] — Adjusted between-group difference in the percentage of participants

45. Secondary Outcome: Number of Participants With a Dental Visit
Description: Child receives a dental screen at least once in first 24 months
Time Frame: Within 24 months after index birth; Medicaid claims and dental records
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 1096 | 509
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 1.7, 95% CI 2-sided [-1.0 to 4.5] — Adjusted between-group difference in the percentage of participants

46. Secondary Outcome: Number of Participants With Fluoride Treatment
Description: Share with recommended fluoride treatments received by child
Time Frame: Within 24 months after index birth; Medicaid claims and dental records
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 1146 | 570
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.2, 95% CI 2-sided [-2.6 to 3.1] — Adjusted between-group difference in the percentage of participants

47. Secondary Outcome: Number of Participants With an Inter-birth Interval of < 24 Months
Description: Having a subsequent birth within the first 24 months of the index birth
Time Frame: Within 24 months after index birth; vital records
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 474 | 244
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -0.3, 95% CI 2-sided [-2.4 to 1.7] — Adjusted between-group difference in the percentage of participants

48. Secondary Outcome: Number of Participants With an Inter-birth Interval of < 15 Months
Description: Having a subsequent birth within the first 15 months of the index birth
Time Frame: Within 15 months after index birth; vital records
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 148 | 85
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -0.7, 95% CI 2-sided [-1.9 to 0.6] — Adjusted between-group difference in the percentage of participants

49. Secondary Outcome: Inter-birth Interval
Description: Continuous measure of inter-birth interval
Time Frame: 60 months after index birth; vital records
Reporting Status: Not Posted, anticipated posting 2027-06

50. Secondary Outcome: Number of Participants With a Family Planning Visit (6 Weeks)
Description: Number of participants who received any family planning-related counseling or service.
Time Frame: Within 6 weeks after index birth; Medicaid claims, hospital discharge
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 1303 | 669
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -1.5, 95% CI 2-sided [-4.3 to 1.3] — Adjusted between-group difference in the percentage of participants

51. Secondary Outcome: Number of Participants Who Received a Highly or Moderately Effective Method of Contraception (6 Weeks)
Description: Received implant, immediate postpartum long-acting reversible contraception (IPP-LARC), long-acting reversible contraception (LARC), or sterilization and moderately effective contraception to include path, ring, diaphragm, injectables and contraceptive pills
Time Frame: Within 6 weeks after index birth; Medicaid claims, hospital discharge
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 1013 | 512
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -0.7, 95% CI 2-sided [-3.4 to 2.0] — Adjusted between-group difference in the percentage of participants

52. Secondary Outcome: Number of Participants Who Received Immediate Postpartum Long-acting Reversible Contraception (6 Weeks)
Description: Number of participants who received immediate postpartum long-acting reversible contraception in first 6 weeks postpartum.
Time Frame: Within 6 weeks after index birth; Medicaid claims, hospital discharge
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 384 | 176
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.8, 95% CI 2-sided [-1.0 to 2.7] — Adjusted between-group difference in the percentage of participants

53. Secondary Outcome: Number of Participants With a Family Planning Visit (1 Year)
Description: Number of participants who received any family planning-related counseling or service in the first year postpartum.
Time Frame: Within 12 months after index birth; Medicaid claims, hospital discharge
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 2378 | 1188
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = -0.4, 95% CI 2-sided [-3.0 to 2.2] — Adjusted between-group difference in the percentage of participants

54. Secondary Outcome: Number of Participants Who Received a Highly or Moderately Effective Method of Contraception (1 Year)
Description: Received implant, IPP-LARC, LARC, or sterilization and moderately effective contraception to include path, ring, diaphragm, injectables and contraceptive pills
Time Frame: Within 12 months after index birth; Medicaid claims, hospital discharge
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 2165 | 1075
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.1, 95% CI 2-sided [-2.6 to 2.9] — Adjusted between-group difference in the percentage of participants

55. Secondary Outcome: Number of Participants Who Received a Postpartum Intrauterine Device Insertion (1 Year)
Description: Number of participants who received a postpartum intrauterine device insertion in first 12 months postpartum.
Time Frame: Within 12 months after index birth; Medicaid claims, hospital discharge
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 476 | 227
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.5, 95% CI 2-sided [-1.5 to 2.6] — Adjusted between-group difference in the percentage of participants

56. Secondary Outcome: Time to First Take-up of Family Planning Counseling or Service
Description: Months from pregnancy to first take up of family planning counseling or service
Time Frame: Within 24 months after index birth; Medicaid claims, hospital discharge
Population: as for outcome 17
Measure: Mean (Standard Error); unit: months
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 2470 | 1229
months | 2 (3.6) | 1.9 (3.3)
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.13, 95% CI 2-sided [-0.1 to 0.37] — Adjusted between-group difference, in months

57. Secondary Outcome: Time to First Take-up of Highly Effective Contraceptive Method
Description: Months from discharge to first take up of highly effective contraceptive method (include implant, IPP-LARC, LARC, or sterilization)
Time Frame: Within 24 months after index birth; Medicaid claims, hospital discharge
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 1016 | 465
months | 2.5 (4.3) | 2.6 (4.5)
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.03, 95% CI 2-sided [-0.45 to 0.5] — Adjusted between-group difference, in months

58. Secondary Outcome: Number of Participants Who Received Supplemental Nutrition Assistance Program (SNAP) or Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) Benefits
Description: Number of participants who received Supplemental Nutrition Assistance Program (SNAP) or Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) benefits during pregnancy.
Time Frame: During index pregnancy, assessed up to 42 weeks; South Carolina Department of Social Services data and birth certificate data respectively
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 2892 | 1408
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 2.1, 95% CI 2-sided [0.3 to 4.0] — Adjusted between-group difference in the percentage of participants

59. Secondary Outcome: Number of Months Receiving SNAP or Temporary Assistance for Needy Families (TANF) Benefits
Description: Total months receiving Supplemental Nutrition Assistance Program or Temporary Assistance for Needy Families
Time Frame: Within 24 months after index birth; South Carolina Department of Social Services data
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of months
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
number of months | 10.4 (9.4) | 9.8 (9.2)
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 0.6, 95% CI 2-sided [0.1 to 1.1] — Adjusted between-group difference, in months

60. Secondary Outcome: Number of Participants With SNAP or TANF Benefit Churn
Description: Receiving Supplemental Nutrition Assistance Program or Temporary Assistance for Needy Families at any time during a given year and having experienced at least one break in participation of four months or less that started and/or ended during the year
Time Frame: Within 24 months after index birth; South Carolina Department of Social Services data
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership | Control
Number analyzed (Participants) | 3295 | 1637
Participants | 382 | 174
Statistical Analysis 1: Comparison: Treatment - Participation in Nurse Family Partnership Nurse-Family Partnership vs Control; Test type: Superiority; Adjusted between-group difference = 1.1, 95% CI 2-sided [-0.7 to 3.0] — Adjusted between-group difference in the percentage of participants

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up (3 years)
Description: We define adverse events in accordance with the Harvard Institutional Review Board (IRB) guidelines as any physical, psychological, social, or economic harms associated with participation in the research. This definition is distinct from that of the National Institutes of Health, which includes all untoward medical occurrences regardless of their relationship to the research. By using the Harvard IRB definition, we report adverse events related to the research or the conduct of the study.
Arm/Group | Treatment - Participation in Nurse Family Partnership | Control
All-Cause Mortality (participants affected / at risk) | 5/3319 | 2/1647
Serious Adverse Events (participants affected / at risk) | 0/3319 | 0/1647
Other Adverse Events (participants affected / at risk) | 0/3319 | 0/1647

LIMITATIONS AND CAVEATS:
The study ended enrollment earlier than planned on March 17, 2020, due to safety concerns arising from the Coronavirus disease 2019 (COVID-19) pandemic. The original plan was to enroll 6,000 mothers (4,000 in the treatment group and 2,000 in the control group) over a four-year period (April 2016-2020), with NFP services provided through the children's second birthday (2016-2022). At the close of enrollment, a total of 5,670 participants had been enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/39/NCT03360539/Prot_001.pdf
  • Statistical Analysis Plan (2025-02-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT03360539/SAP_002.pdf
  • Informed Consent Form (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/39/NCT03360539/ICF_000.pdf